CLINICAL TRIAL: NCT03264820
Title: Study of the Reproducibility of Laser Measurement in the Detection of Digital
Brief Title: Study of the Reproducibility of Laser Measurement in the Detection of Digital Obstructive Arterial Disease (DOAD)
Acronym: REPROLASER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator decision
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC169738
Record Dates: First submitted 2017-07-28; First posted 2017-08-29 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Vascular Diseases
Keywords: digital obstructive arterial disease, DOAD
MeSH Terms: conditions — Vascular Diseases | interventions — Laser-Doppler Flowmetry; Laser Speckle Contrast Imaging; Blood Pressure; Heart Rate

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, non-randomized study 11 healthy volonteer 33 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with scleroderma and potential arterial disease (Experimental): The patients (33) will undergo a medical examination in order to analyse their medical history, parameters and check inclusion and non-inclusion criterions.
  Then will be performed :
  Visit 1 :
  * Biology report * (* Biological evaluation carried out in all healthy subjects and in subjects whose biological check-up dates more than 2 years,+ urinary pregnancy test (if applicable))
  * Laser measurements at the forearm (with laser speckle)
  * Laser measurements at the level of each finger
  * Pain evaluation (EVA)
  * Measurement of blood pressure and heart rate
  * Environmental measures and skin temperature
  Visit 2 :
  * Laser measurements at the level of each finger
  * Pain evaluation (EVA)
  * Measurement of blood pressure and heart rate
  * Environmental measures and skin temperature
  Interventions: Device: Laser Doppler; Device: Laser speckle; Behavioral: pain evaluation; Other: Blood pressure and heart rate
- Healthy volunteers (Experimental): The healthy volunteers (11) will undergo :
  Visit 1 :
  * Biology report (+ urinary pregnancy test (if applicable))
  * Laser measurements at the forearm (with laser speckle)
  * Laser measurements at the level of each finger
  * Pain evaluation (EVA)
  * Measurement of blood pressure and heart rate
  * Environmental measures and skin temperature
  Visit 2 :
  * Laser measurements at the level of each finger
  * Pain evaluation (EVA)
  * Measurement of blood pressure and heart rate
  * Environmental measures and skin temperature
  Interventions: Device: Laser Doppler; Device: Laser speckle; Behavioral: pain evaluation; Other: Blood pressure and heart rate

INTERVENTIONS:
Device: Laser Doppler — - Laser measurements at the level of each finger at 47 °C and at ambient temperature
Device: Laser speckle — - Laser measurements at the forearm
Behavioral: pain evaluation — Visual scale assesment pain
Other: Blood pressure and heart rate — Measurement of blood pressure and heart rate

SUMMARY:
At the digital level, the diagnosis of obstructive arteriopathy is very difficult in the absence of ulcer or of true ischemic signs, and the arteriography, which is an examination to inject an intra-arterial contrast agent, is the reference measure.

The measure by "Laser Doppler" uses a monochromatic light (laser) to measure the concentration as well as the speed of travel of red blood cells in the skin and deduct the cutaneous blood flow.

The great advantage of this technique is that it is non-invasive, inexpensive and can be performed during a consultation. The patient can therefore be briefly informed of the benign (functional) or organic origin of his disorders.

DETAILED DESCRIPTION:
In the systematic sclérodermie, 15 to 25 % of the patients suffer from active digital ulcers and 35 to 50 % of the patients will make a digital ulcer. These digital ulcers are in touch with an obstructive digital arteriopathy, that is arterial hurts modifying the arterial flow. It thus seems interesting to have diagnostic tools allowing to make the diagnosis in particular upstream to the appearance of ulcers. At present, the digital pressures can be used.

At the digital level, the diagnosis of obstructive arteriopathy is very difficult in the absence of ulcer or of true ischemic signs, and the arteriography, which is an examination to inject an intra-arterial contrast agent, is the reference measure.

For this study, the investigator shall use the Laser doppler PeriFlux 5000 system (Perimed, Jarfalla, Sweden - List IIa) who is regularly used in clinical routine and who has a marking IT for the recording of the blood flow at the cutaneous level for the measures of blood pressure in particular (measures of pressures in the big toe and in the fingers).

The measure by "Laser Doppler" uses a monochromatic light (laser) to measure the concentration as well as the speed of travel of red blood cells in the skin and deduct the cutaneous blood flow. This material is used in this project because the investigators have already highlighted with this one that the detection of an obstructive digital arteriopathy was excellent.

Given the invasive and costly nature of arteriography, it is only very rarely performed. Moreover, this can not be carried out during a simple consultation.

Nevertheless, it is important for the patient and the practitioner to determine whether the digital symptoms are related to benign vasomotor phenomena or to a real digital arterial disease. The therapeutic management is different.

ELIGIBILITY:
Inclusion Criteria:

* Patients :
* Adult 18 years of age or older;
* Woman of childbearing age under effective contraception for 1 month (IUD, pill, implant);
* Presenting scleroderma;
* Able to understand the objectives of the study and its constraints;
* Affiliated to social security;
* Having given free, informed and written consent

Healthy volunteers:

* Adult 18 years of age or older;
* Woman of childbearing age under effective contraception for 1 month (IUD, pill, implant);
* Not presenting and showing no Raynaud syndrome and / or digital ulceration;
* Able to understand the objectives of the study and its constraints;
* Affiliated to social security;
* Having given free, informed and written consent

Exclusion Criteria for healthy volunteers and patients

* subjects in periods of exclusion relating to another biomedical study;
* subjects with declared pregnancy;
* breastfeeding patients
* having an allergy to adhesives;
* protected majorities (safeguard of justice, curatorship, guardianship) and persons deprived of their liberty
* hospitalized in a health or social institution for any reason other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Reproducibility | Change between baseline and day 15 measure
  Change of Doppler laser measurement in subjects with scleroderma.

SECONDARY OUTCOMES:
Blood flow signal characteristics | Change between baseline and day 15 measure
  To study changes in the signature of the blood flow signal between healthy subjects and subjects with scleroderma.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MAHE, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes _ Service de radiologie et imagerie médicale, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided
It is indicated in the consent of the patient that his data may be transferred to other searchers in France or abroad in the future

REFERENCES:
- [Derived] Omarjee L, Metairie A, Tueguem Moyo T, Pabic EL, Jego P, Lescoat A, Mahe G. Performance of finger systolic blood pressure measurement to detect digital occlusive arterial disease in systemic sclerosis. Rheumatology (Oxford). 2022 Mar 2;61(3):1115-1122. doi: 10.1093/rheumatology/keab497. PMID 34142126